CLINICAL TRIAL: NCT01389791
Title: MgSO4 Combined With Rocuronium Priming
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kim Mihyun, full instructor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mg priming
Record Dates: First submitted 2011-05-26; First posted 2011-07-08 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Muscle Relaxation
Keywords: muscle relaxation; magnesium sulfate; rocuronium
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Roc (No Intervention): Patients in this group receive neither MgSO4 nor priming dose of rocuronium.
- priming (Active Comparator): patients in this group receive 0.06mg/kg of rocuronium before 0.54mg/kg of rocuronium.
  Interventions: Drug: priming
- Mg&priming (Experimental): Patients in this group receive MgSO4 50mg/kg and 0.06mg/kg of rocuronium before administration of 0.54mg/kg of rocuronium.
  Interventions: Drug: magnesium sulfate and priming
- MgSO4 (Active Comparator): Patients in this group receive intravenous MgSO4 before administration of rocuronium.
  Interventions: Drug: magnesium sulfate

INTERVENTIONS:
Drug: magnesium sulfate — Patients in this group receive intravenous MgSO4 50mg/kg before administration of rocuronium (induction dose).
  Other Names: MgSO4
  Arms: MgSO4
Drug: priming — Patients in this group receive 0.06mg/kg of rocuronium before administration of 0.54mg/kg of rocuronium.
  Other Names: rocuronium-priming
  Arms: priming
Drug: magnesium sulfate and priming — Patients in this group receive MgSO4 50mg/kg and 0.06mg/kg of rocuronium before administration of 0.54mg/kg of rocuronium.
  Other Names: MgSO4 & priming
  Arms: Mg&priming

SUMMARY:
Priming with either rocuronium or MgSO4 is known to accelerate the effect of rocuronium on muscle relaxation. The purpose of this study is to define the effect of MgSO4 on the rocuronium-priming.

DETAILED DESCRIPTION:
Acceleration of muscle relaxation is beneficial in rapid-sequence intubation. If MgSO4 combined with priming is efficient in accelerating muscle relaxation, it would be an interesting alternative to rapid-sequence intubation.

ELIGIBILITY:
Inclusion Criteria:

* patients of ASA Ⅰ-Ⅱ
* aged 18~65
* scheduled to undergo elective surgery under general anesthesia

Exclusion Criteria:

* risk of pulmonary aspiration
* anticipated airway difficulty
* reactive airway disease
* allergic to study drugs
* neuromuscular / cardiovascular/ renal/ hepatic disease
* atrioventricular conduction disturbance
* BMI < 18.5 or > 24.9
* chronic treatment with calcium channel blocker
* medications which affect muscle relaxation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
time from injection of induction dose of rocuronium until 95% depression of TOF | time from injection of induction dose of rocuronium until 95% depression of TOF, upto 5 min

SECONDARY OUTCOMES:
rocuronium duration | time from injection of induction dose of rocuronium until train-of-four count reaches two.
  time from injection of induction dose of rocuronium until train-of-four count reaches two.
intubating condition | time from injection of induction dose of rocuronium until tracheal intubation.
  rapid sesequence intubation condition is evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Sanghwan Do, M.D., PH.D., Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul national university Bundang hospital, Seongnam, Kyoung-ki-do, South Korea